CLINICAL TRIAL: NCT03765983
Title: Phase II Trial of GDC-0084 in Combination With Trastuzumab for Patients With HER2-Positive Breast Cancer Brain Metastases
Brief Title: GDC-0084 in Combination With Trastuzumab for Patients With HER2-Positive Breast Cancer Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: participants are no longer being examined or receiving intervention
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Kazia Therapeutics Limited (Industry)
Responsible Party: Principal Investigator, Jose Pablo Leone, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-516
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; GDC-0084

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: single-arm, two stage, phase II cohort (Experimental): GDC-0084 45 mg administered orally once daily Trastuzumab administered at a dose of 8 mg/kg intravenously (IV) loading dose; followed by 6 mg/kg IV every 3 weeks thereafter
  Interventions: Drug: Trastuzumab; Drug: GDC-0084
- Cohort B: a pre-surgical window cohort (Experimental): GDC-0084 45 mg administered orally once daily Trastuzumab administered at a dose of 8 mg/kg intravenously (IV) loading dose; followed by 6 mg/kg IV every 3 weeks thereafter Surgical brain metastasis resection
  Interventions: Drug: Trastuzumab; Drug: GDC-0084

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab is called a "targeted therapy" because it works by attaching itself to specific receptors on the surface of breast cancer cells, known as HER2 receptors. When targeted therapies attach to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the immune system
Drug: GDC-0084 — GDC-0084 has been shown to stop the activity of a protein called PI3-kinase. This action blocks a pathway in the body that cancer cells commonly use to grow and divide

SUMMARY:
This research study is studying a drug called GDC-0084 as a possible treatment for HER2-Positive Breast Cancer.

The drugs involved in this study are:

* GDC-0084
* Trastuzumab (Herceptin®)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved GDC-0084 as a treatment for any disease.

Trastuzumab is a targeted therapy approved by the FDA to be used alone or in combination with a chemotherapy drug to treat HER2-positive metastatic breast cancer.

GDC-0084 has been shown to stop the activity of a protein called PI3-kinase. This action blocks a pathway in the body that cancer cells commonly use to grow and divide.

Trastuzumab is called a "targeted therapy" because it works by attaching itself to specific receptors on the surface of breast cancer cells, known as HER2 receptors. When targeted therapies attach to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the immune system. This process allows trastuzumab to help slow or stop the growth of the breast cancer.

In this research study, the investigators are looking to see how your cancer responds to the combination of GDC-0084 and Trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* At least one measurable CNS metastasis, defined as ≥ 10 mm in at least one dimension.
* Unequivocal evidence of new and/or progressive brain metastases, and at least one of the following scenarios:

  * Treated with SRS or surgery with residual un-treated lesions remaining. Such participants are eligible for immediate enrollment on this study providing that at least one untreated lesion is measurable
  * Participants who have had prior WBRT and/or SRS and then whose lesions have subsequently progressed or who have new lesions are also eligible. In this case, lesions which have been treated with SRS may be considered as target lesions if there is unequivocal evidence, in the opinion of the treating physician, of progression following SRS.
  * Participants who have not previously been treated with cranial radiation (e.g., WBRT or SRS) are eligible to enter the study, but such participants must be asymptomatic from their CNS metastases and not requiring corticosteroids for symptom control.
  * Participants who present with systemic stable/absent or progressive disease are eligible to this trial, as long as they fulfill one of the above criteria.

Cohort B:

* New and/or progressive brain metastasis(es) with clinical indication for resection.
* All Cohorts:
* Pathologically confirmed HER2-positive MBC by local laboratory with the following requirements: HER2 overexpressed or amplified (immunohistochemistry of 3+ or HER2 gene amplification by in situ hybridization with a ratio of HER2-gene signals to centromere 17 signals ≥ 2.0 or average HER2 copy number ≥ 6.0 signals/cells).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
* Stable or decreasing corticosteroid dose for at least 7 days prior to initiation of treatment.
* Concurrent administration of other anti-cancer therapy during the course of this study is not allowed. Note that concurrent use of supportive care medications (e.g. anti-resorptive agents, pain medications) is allowed.
* The participant is ≥18 years old.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/μl
  * Platelets ≥75,000/μl
  * Hemoglobin ≥9 g/dL
  * Total bilirubin ≤1.5mg/dL (upper limit of normal) except subject with documented Gilbert's syndrome (≤5 x ULN) or liver metastasis, who must have a baseline total bilirubin ≤3.0 mg/dL;
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN OR ≤ 5.0 × institutional ULN for patients with documented liver metastases.
  * Serum creatinine ≤ 1.5 mg/dL (or glomerular filtration rate ≥ 30 ml/min as determined by the Cockcroft-Gault equation)
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 8 days of initiating protocol therapy.
* The effects of GDC-0084 on the developing human fetus are unknown and radiotherapy has known teratogenic effects so women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 7 months after completion of Trastuzumab administration per recommendations from the Trastuzumab package insert.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
* Participant must be able to swallow and retain oral medication.

Exclusion Criteria:

* Visceral crisis or impending visceral crisis at time of screening.
* CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement).
* Known leptomeningeal metastases [Defined as positive CSF cytology and/or unequivocal radiological evidence of clinically significant leptomeningeal involvement. CSF sampling is not required in the absence of suggestive symptoms to exclude leptomeningeal involvement].
* Patients with known contraindication to MRI (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity, hypersensitivity, etc.). However, head CT with contrast may be used in place of MRI at baseline and throughout the trial if MRI is contraindicated and a participant's brain metastases are clearly measurable by head CT.
* Chemotherapy or targeted therapy within 14 days prior to initiation of protocol therapy. No washout is required for trastuzumab.
* Has received prior therapy with a PI3K or mTOR inhibitor.
* No washout is required for endocrine therapy. If a patient has been on ovarian suppression for at least 28 days prior to initiation of study treatment, continuation of ovarian suppression is permitted on protocol. Starting a new endocrine therapy during protocol therapy is not permitted.
* Current use or history of receiving a non-approved, investigational treatment within 14 days prior to initiation of protocol therapy.
* Subjects with a history of hypersensitivity to compounds of similar biologic composition to GDC-0084 or any constituent of the product.
* The subject has an uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus (DM), gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, or severe malnutrition. If a participant has controlled DM but is unable to monitor blood sugars at home, they will be excluded from the trial.
* The subject is pregnant or breast-feeding.
* No active, second potentially life-threatening cancer.
* Has had major surgery within 21 days before initiation of protocol therapy.
* Active infection requiring IV antibiotics at the time of protocol therapy initiation.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest.
* Known intolerance to trastuzumab.
* QT interval time of ≥ 470 msec.
* Participants receiving any medications or substances that are strong inhibitors or strong inducers of CYP3A4 are ineligible. Should a participant be taking one of these agents and is able to discontinue the therapy or switch to a different agent, no washout will be required prior to starting study medication. Please see Appendix M for the list of medications. Corticosteroids, which are weak CYP3A4 inducers are allowed. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate in the CNS | 2 years
  ORR in the CNS according to response assessment in neuro-oncology-brain metastases (RANO-BM) criteria
To evaluate the correlation between inhibition of p-4EBP1 in resected brain tumor tissue and intracranial response in the corresponding patient-derived xenograft (PDX) models of BCBM | 2 Years
  to correlate on-treatment p4EBP1 levels in the resected brain tumor tissue collected from patients to intracranial response to GDC-0084/trastuzumab and survival in the PDX model generated from the same patient

SECONDARY OUTCOMES:
CBR | 18 and 24 weeks
  rate of patients with clinical benefit at 18 and 24 weeks
DOR | 2 years
  to measure the duration of response in the CNS
Objective extra-CNS response rates | 2 years
  the rate of patients who have an objective response outside of the CNS
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  to evaluate the number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Progression Free Survival | 2 years
  measured by RANO-BM and RECIST 1.1
Overall Survival | 2 years
  to evaluate overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jose P Leone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor-Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than one year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor-Investigator or designee].